CLINICAL TRIAL: NCT02195661
Title: The Role of Melatonin in the Effective Attainment of Sleep Electroencephalograms (EEG) in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Jo M Wilmshurst, Professor Jo Wilmshurst, University of Cape Town
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 070/2014
Record Dates: First submitted 2014-07-16; First posted 2014-07-21 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Epilepsy; Electroencephalogram; Children; Sedation
Keywords: Epilepsy; Electroencephalogram; children; sedation
MeSH Terms: conditions — Epilepsy | interventions — Melatonin; Chloral Hydrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melatonin sleep EEG induced group (Active Comparator): All children who were referred to the neurophysiology department who were either unable to keep still for their EEG, or required a sleep EEG as part of their epilepsy "work-up" and whose caregivers agreed to the administering of sedation with melatonin. Melatonin by mouth (3mg for children < 15kg, 6mg for those > 15kg) 1 hour before the scheduled EEG by the unit nurse. Children who can swallow the capsules directly, those who cannot are given the contents of the powder in the capsule mixed in a few millilitres of water. If the child fails to fall asleep within one hour of administration of the melatonin then a second dose 3mg is given) .
  Interventions: Dietary Supplement: Melatonin
- Comparison group for children sedated using previous practice (Other): Since the choral hydrate had been withdrawn a direct comparison group was not possible. However a study performed the previous year in the department measured a several parallel useful outcomes. This study had addressed the usefulness of electroencephalograms in a South African population. A proportion of this group screened in 2012 in our unit underwent sleep studies, sedated with chloral (n=22). These patients were drawn from the same regional pool, with the same disease demographics, and the same sleep deprivation and procedural techniques to the current group. This group was screened for several common denominators to the current study themes, and comparison will be made between these, namely the proportion of patients with successful attainment of sleep studies, the proportion of studies with excessive artifact (precluding interpretation) and the usefulness of the data attained detailing whether the studies were able to assist or alter patient management.
  Interventions: Drug: Chloral Hydrate

INTERVENTIONS:
Dietary Supplement: Melatonin
  Arms: Melatonin sleep EEG induced group
Drug: Chloral Hydrate
  Arms: Comparison group for children sedated using previous practice

SUMMARY:
This study aims to determine the safety and effectiveness of oral melatonin as natural inducer of sleep to acquire useful EEGs in South African children following its introduction as the main agent used in the Neurophysiology department at Red Cross Children's Hospital. This is an observational retrospective study.

ELIGIBILITY:
Inclusion Criteria:

* All children who were referred to the neurophysiology department who were either unable to keep still for their EEG, or required a sleep EEG as part of their epilepsy "work-up" and whose caregivers agreed to the administering of sedation with melatonin.

Exclusion Criteria:

* Those children undergoing prolonged EEG monitoring (telemetry) or within 24 hours of status epilepticus (prolonged or cluster of seizures).
* Those children are not sedated as natural sleep is always attained with the prolonged monitoring studies, and for those with status epilepticus, there is usually evidence on the EEG of alteration secondary to the effects of status, and the medications administered to control the presenting event.
* Any child deemed to unwell to undergo a non-emergency procedure.
* Any child already receiving anticoagulant medications.
* Any caregiver who deferred sedation for their child was also excluded from the study and in the unit the procedure attempted without sedation.

Ages: 6 Months to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 194 (Actual)
Dates: Start 2014-04; Primary Completion 2017-09 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of melatonin to induce sleep for EEG studies | 6 months
  Successful attainment of EEG (in comparison to the unit's previous success rate)(Definition: "successful attainment of EEG" = completed sleep EEG, without excessive artefact enabling an comprehensive report to be generated in a child who undergoes the procedure without evidence of adverse drug reactions)

SECONDARY OUTCOMES:
Breakdown data from the successful EEGs - | 6 months
  Yield in terms of EEG abnormalities - number of abnormal studies, number of studies yielding outcomes which will alter patient management

OTHER OUTCOMES:
Comparison of EEGs performed under melatonin sedation compared to previous unit protocol | 6 months
  To compare the EEG recordings in comparison to a historical group of age matched recordings sedated with chloral and to establish if the outcomes achieved are in line with the previous unit practice.

CONTACTS AND LOCATIONS:
Locations (1):
- Red Cross War Memorial Children's Hospital, Cape Town, Western Cape, South Africa

REFERENCES:
- [Background] Ibekwe R, Jeaven L, Wilmshurst JM. The role of melatonin to attain electroencephalograms in children in a sub-Saharan African setting. Seizure. 2017 Oct;51:87-94. doi: 10.1016/j.seizure.2017.08.002. Epub 2017 Aug 12. PMID 28826048